CLINICAL TRIAL: NCT02298530
Title: A Study to Determine the Acute Effects of a Tea Component on Blood Pressure and Mental Stress Challenge
Brief Title: Tea Components, Mental Stress and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REF-BEV-1803
Record Dates: First submitted 2014-11-12; First posted 2014-11-24 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
MeSH Terms: interventions — theanine; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination of caffeine and theanine (Experimental): 250 mg caffeine + 200 mg theanine
  Interventions: Other: Combination of caffeine and theanine
- Caffeine (Placebo Comparator): 250 mg caffeine
  Interventions: Other: Caffeine

INTERVENTIONS:
Other: Combination of caffeine and theanine — Beverage containing caffeine and theanine
  Arms: Combination of caffeine and theanine
Other: Caffeine — Beverage containing caffeine
  Arms: Caffeine

SUMMARY:
Assess the effects of adding theanine to a caffeinated beverage on changes in blood pressure during acute mental stress.

DETAILED DESCRIPTION:
Caffeine and (mental) stress can increase blood pressure. In a typical everyday and/or work environment they commonly coincide. Tea has the reputation of being a relaxing drink. L-theanine is an amino acid found almost exclusively in tea. In a previous study it was shown that caffeine increased blood pressure, while theanine antagonised these effects. In the current study the effect of theanine to a placebo on blood pressure are directly compared.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males and females
* Women taking the contraceptive pill
* 18-45 years of age
* BMI 20-30 kg/m2
* Normal or corrected vision
* Low caffeine consumers (<100mg/day)
* Non smokers and having been a non-smoker for > 6 months
* Fluent English
* Normotensive (>90/60 <140/90 mmHg)

Exclusion Criteria:

* Significant current or medical history of cardiovascular disease
* Low or high STAI trait score in the opinion of the PI
* Known sensitivity to caffeine or theanine
* Colour blindness
* Alcohol consumption above 14/21 units female/male resp. per week
* Weight loss diet > 10% of bodyweight in the previous year
* Anyone with a dependency on PI or staff of Department of Epidemiology and Public Health or being an employee of Unilever
* Reported participation in another biomedical study < 3 months before screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure during stress | Between 30-45 minutes after test product intake
  Systolic blood pressure during acute mental stress

SECONDARY OUTCOMES:
Diastolic blood pressure during stress | Between 30-45 minutes after test product intake
  Diastolic blood pressure during acute mental stress
Systolic blood pressure after stress | Between 45-60 minutes after test product intake
  Systolic blood pressure immediately after acute mental stress
Diastolic blood pressure after stress | Between 45-60 minutes after test product intake
  Diastolic blood pressure immediately after acute mental stress
STAI before and immediately after stress | -15 and 45 relative to test product intake
  Self-reported mental state: State-Trait Anxiety Inventory
UWIST before and immediately after stress | -10, 45 minutes relative to test product intake
  Self-reported mental state: University Of Wales Institute of Science and Technology mood adjective questionnaire

OTHER OUTCOMES:
Cortisol in saliva before and immediately after stress | -5, 45 min relative to test product intake
  Concentration of cortisol in saliva
Heart rate during stress | Between 30-45 minutes after test product intake
  Heart rate during acute mental stress
Heart rate after stress | Between 45-60 minutes after test product intake
  Heart rate immediately after acute mental stress
Heart rate variability during stress | Between 30-45 minutes after test product intake
  Heart rate variability during acute mental stress
Heart rate variability after stress | Between 45-60 minutes after test product intake
  Heart rate variability immediately after acute mental stress
Performance STROOP | Between 30-45 minutes after test product intake
  Task performance on STROOP task
Performance mirror tracing | Between 30-45 minutes after test product intake
  Task performance on mirror tracing task
Systolic blood pressure, free living phase | Between 80-270 minutes after test product intake
  Ambulatory systolic blood pressure during free living phase
Diastolic blood pressure, free living phase | Between 80-270 minutes after test product intake
  Ambulatory diastolic blood pressure during free living phase
Cortisol, free living phase | 140, 200 and 260 minutes after test product intake
  Concentration of cortisol in saliva during free living phase
STAI, free living phase | 140, 200 and 260 minutes after test product intake
  Self-reported mental state: State-Trait Anxiety Inventory during free living phase
UWIST, free living phase | 140, 200 and 260 minutes after test product intake
  Self-reported mental state: University Of Wales Institute of Science and Technology) mood adjective questionnaire during free living phase
Pulse pressure during stress | Between 30-45 minutes after test product intake
  Mean pulse pressure during mental stress
Pulse pressure after stress | Between 45-60 minutes after test product intake
  Mean pulse pressure after acute mental stress
Mental wellbeing | 7 consecutive days prior to the lab sessions
  Mental well being as assessed by on line survey an each evening during the 7 day period the accelerometer is worn.
Physical activity | 7 consecutive days prior to the lab sessions
  Habitual patterns in physical activity as measured by accelerometer
STAI screening | Screening
  State-Trait Anxiety Inventory (STAI) - Trait version, covariate
CES-D | Screening
  Center for Epidemiologic Studies Depression scale, covariate
CISS | Screening
  CISS coping scale, covariate
loneliness | Screening
  UCLA loneliness scale, covariate
Perceived stress | Screening
  Perceived Stress Scale, covariate

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hamer, Dr, Principal Investigator — UCL, Epidemiology & Public Health, London
Locations (1):
- University College London, London, United Kingdom